CLINICAL TRIAL: NCT05375279
Title: A PILOT Study on Labial Salivary Gland Biopsy Potentially to Replace Endomyocardial Biopsy in the Diagnosis of Cardiac Transthyretin Amyloidosis
Brief Title: A PILOT Study on LSGB vs EMB in the Diagnosis of Cardiac Transthyretin Amyloidosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Unity Health Toronto (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Gordon Moe, Investigator, Unity Health Toronto
Other Study IDs: 70095215
Record Dates: First submitted 2022-05-10; First posted 2022-05-16 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Amyloidosis
Keywords: Amyloidosis; Cardiomyopathy
MeSH Terms: conditions — Amyloidosis; Cardiomyopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LSGB vs EMB: Patients who already underwent EMB within the last six months with confirmed Amyloid Transthyretin -wild type (ATTRwT) will undergo LSGB.
  Interventions: Procedure: Lip Salivary Gland Biopsy

INTERVENTIONS:
Procedure: Lip Salivary Gland Biopsy — Obtaining few salivary glands from the partipants' lip that will be studied using the Congo Red staining method.

SUMMARY:
Transthyretin (TTR) is a plasma protein mainly synthesized in the liver, recognized as a transporter of thyroxine and retinol-binding protein. Unstable changes in two types of TTR (wild type or variant) become misfolded, aggregate, and ultimately forms amyloid fibrils. Amyloid Transthyretin Cardiac amyloidosis (ATTR-CA) is an infiltrative cardiomyopathy caused by extracellular deposition of insoluble transthyretin (TTR) amyloid fibrils in the heart muscle. Cardiac amyloidosis (CA) has been recognized as a common cause of heart failure with preserved ejection fraction (HFpEF) among elderly persons, with increasing incidence.

There are different ways of diagnosing ATTR-CA. These include cardiac magnetic resonance imaging, nuclear scintigraphy, and tissue biopsy, the gold standard. Tissues biopsy extracted from the adipose, lip salivary gland (LSG), and heart muscle (endomyocardial biopsy or EMB).

Tissue diagnosis is the prerequisite of provincial support of the disease-modifying agent. However, with the convenience, ease, less risk of bleeding, and high sensitivity, LSG may offer an alternative to the more invasive EMB to diagnose suspected CA.

To test the hypothesis that LSGB can replace EMB in tissue diagnosis of ATTR-CM.

This Pilot study is designed to evaluate two invasive diagnostic methodologies: LSGB and the EMB. A total of 20 patients who underwent EMB within the last six months with confirmed Amyloid Transthyretin -wild type (ATTRwT) will be invited to participate. In addition, patients who signed the informed consent form will be scheduled for LSGB within two weeks.

DETAILED DESCRIPTION:
We propose broad eligibility criteria to increase the generalizability and feasibility of the proposed study. Patients who are confirmed diagnosis of Amyloid Transthyretin Cardiomyopathy - wild type (ATTRwt) through Echocardiography, Cardiac Magnetic Resonance Imaging, pyrophosphate scan, and genetic testing and had an endomyocardial biopsy (or will undergo endomyocardial biopsy) are eligible to participate in the study.The exclusion criteria are predominantly patients who had negative amyloid deposits in the endomyocardial biopsy. There are no exclusions based on gender, race or ethnicity in this trial.

LSG biopsy will be performed under local anesthesia (2% lidocaine). The lip will be everted, and a 3 to 4 mm longitudinal incision will be made in the labial mucosa in front of the mandibular canine tooth. Three minor salivary glands will be exposed and removed. No silk suture will be used. [18] The LSG specimen will match the EMB specimen. LSG biopsy tissues will be studied using the method of Congo red stain.[18] The participants will be scheduled for LSGB at the London Health Sciences Centre within two weeks of signing the informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are confirmed diagnosis of Amyloid Transthyretin Cardiomyopathy - wild type (ATTRwt) through Echocardiography, Cardiac Magnetic Resonance Imaging, pyrophosphate scan, and genetic testing and had an endomyocardial biopsy (or will undergo endomyocardial biopsy).

Exclusion Criteria:

* Patients who had negative amyloid deposits in the endomyocardial biopsy.

Ages: 18 Years to 96 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are confirmed diagnosis of Amyloid Transthyretin Cardiomyopathy - wild type (ATTRwt) through Echocardiography, Cardiac Magnetic Resonance Imaging, pyrophosphate scan, and genetic testing and had an endomyocardial biopsy (or will undergo endomyocardial biopsy).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-06-15 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
LSG biopsy with positive amyloid deposits will be observed in a higher proportion in patients with positive EMB. | 6 months
  Proportions of patients who will test positive and negative will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Gordon W Moe, MD, FRCPC, FACC, Principal Investigator — Unity Health Toronto
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No